CLINICAL TRIAL: NCT06427850
Title: Effect of Topical Tranexamic Acid on Postoperative Drainage in Minimally Invasive Transforaminal Lumbar Interbody Fusion (MI-TLIF): A Randomized Controlled Trial
Brief Title: Effect of Topical Tranexamic Acid on Postoperative Drainage in Minimally Invasive Transforaminal Lumbar Interbody Fusion (MI-TLIF)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thanawan Longsuwan (Other)
Responsible Party: Sponsor-Investigator, Thanawan Longsuwan, Doctor, Ramathibodi Hospital
Organization: Ramathibodi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123678
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Degenerative Spine Diseases; Surgical Wound
Keywords: Degenerative spine diseases; Surgical wound; Tranexamic acid (TXA)
MeSH Terms: conditions — Surgical Wound | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical tranexamic acid (TXA) injection (Experimental): receive an injection of topical tranexamic acid (TXA) into the surgical site
  Interventions: Drug: Tranexamic acid
- Placebo group (Placebo Comparator): receive an injection Normal saline into the surgical site
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic acid — receive an injection of Tranexamic acid into the surgical site
  Arms: Topical tranexamic acid (TXA) injection
Drug: Normal saline — receive an injection of Normal saline into the surgical site
  Arms: Placebo group

SUMMARY:
The randomized controlled study which compare the efficacy outcomes (reducing blood loss and drainage output in patients) in patients undergoing single-level minimally invasive transforaminal lumbar interbody fusion (MI-TLIF) and received topical tranexamic acid injection in the surgical site to those who received placebo injection.

DETAILED DESCRIPTION:
Detail : Randomization of Patients for intra-surgical site topical tranexamic acid injection

Objective : To compare the efficacy of topical tranexamic acid (TXA) injection into the surgical wound versus placebo injection in reducing blood loss and drainage output in patients undergoing single-level minimally invasive transforaminal lumbar interbody fusion (MI-TLIF) surgery.

Methods:

Patient: Patients with degenerative spine conditions undergoing single-level MI-TLIF surgery, who received treatment at Ramathibodi Hospital and Chakri Naruebodindra Medical Institute from 2024 to 2027.

Randomization : Patients will be randomly by various block randomization (1:1) was performed using STATA 16.0 to ensure that the two groups were comparable in size and that the sequence of randomization was unpredictable.

Intervention :

Group 1 : Patients in this group will receive an injection of topical tranexamic acid (TXA) into the surgical site(50mg/ml) 10 ml after wound exposure and after wound decompression.

Group 2: Patients in this group will receive a placebo injection (Normal saline 10 ml) into the surgical site after wound exposure and after wound decompression.

Allocation Concealment :

A central randomization service will prepare sealed envelopes labeled with sequence numbers corresponding to the sample size. This method decreasing selection bias in assigning participants to the treatment groups. The envelopes were opened and equipment prepared after anesthesia was administered and before the surgeon began the incision.

Blinding :

The study participants and assessors will be blinded to treatment allocation. The surgeons were blinded by clear fluid as same in 2 groups but if tranexamic acid can be effective to decrease blood loss in intraoperation. So we cannot controlled blinding surgeons.

Primary outcome measurement: postoperative drainage (ml)

Secondary outcome measurement:

calculated total blood loss, intraoperative blood loss, blood transfusion rate, duration of drain maintenance, length of hospital stay, complication of tranexamic acid (TXA) and surgery.

Statistical Analysis:

Demographic Analysis :

For continuous data reported as Mean and Standard Deviation (S.D.) and analyzed by Independent t-test or Mann-Whitney U test.

For categorical data reported as Percentages and analyzed by Chi-square test.

Compare the results of the study:

Postoperative drainage (ml),calculated total blood loss (ml), intraoperative blood loss (mL) , duration of drain maintenance (day), length of hospital stay (day)were report to Mean and Standard Deviation (S.D.) analyzed by Independent t-test or Mann-Whitney U test for continuous data.

Complication of tranexamic acid (TXA) and surgery(%), blood transfusion rate (%) were reported to Percentages and analyzed by Chi-square test. Use STATA 16.0 software for statistical calculations.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80 years old
* Degenerative spine problems including spinal stenosis, disc degeneration, spondylolithesis that indicated for single level MI-TLIF

Exclusion Criteria:

* Revision surgery
* Patients who had high risk of complication from TXA
* History of seizure, PE, DVT, thromboembolic episode
* History of TXA allergy
* Patients who had high risk for bleeding
* U/D : CKD stage more than IIIb (GFR< 45 ml/min/1.73m2), hepatic disease, bleeding disorder
* On anticoagulation drug or antiplatelet drug in 7 days before surgery
* Abnormal coagulation profile (INR > 1.5) or CBC (platelet < 100000)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
postoperative drainage (mL) | 120 hours
  Fluid drainage after operation

SECONDARY OUTCOMES:
calculated total blood loss (mL) | 120 hours
  calculated total blood loss by Gross formular
intraoperative blood loss (mL) | Intraoperative time
  Evaluated by anesthesiologists
duration of drain maintenance (day) | 120 hours
  Duration time of drain insertion to off drain
length of hospital stay (day) | 120 hours
  Duration time of patients stay in hospital
complication of tranexamic acid (TXA) and surgery(%) | 120 hours
  The patients who had complication from tranexamic acid (TXA) and surgery in each group

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ravindra VM, Senglaub SS, Rattani A, Dewan MC, Hartl R, Bisson E, Park KB, Shrime MG. Degenerative Lumbar Spine Disease: Estimating Global Incidence and Worldwide Volume. Global Spine J. 2018 Dec;8(8):784-794. doi: 10.1177/2192568218770769. Epub 2018 Apr 24. PMID 30560029
- [Background] Atlas SJ, Keller RB, Wu YA, Deyo RA, Singer DE. Long-term outcomes of surgical and nonsurgical management of lumbar spinal stenosis: 8 to 10 year results from the maine lumbar spine study. Spine (Phila Pa 1976). 2005 Apr 15;30(8):936-43. doi: 10.1097/01.brs.0000158953.57966.c0. PMID 15834339
- [Background] Harms JG, Jeszenszky D. Die posteriore, lumbale, interkorporelle Fusion in unilateraler transforaminaler Technik. Oper Orthop Traumatol. 1998 Jun;10(2):90-102. doi: 10.1007/s00064-006-0112-7. No abstract available. German. PMID 17332991
- [Background] Holly LT, Schwender JD, Rouben DP, Foley KT. Minimally invasive transforaminal lumbar interbody fusion: indications, technique, and complications. Neurosurg Focus. 2006 Mar 15;20(3):E6. doi: 10.3171/foc.2006.20.3.7. PMID 16599422
- [Background] Moskowitz A. Transforaminal lumbar interbody fusion. Orthop Clin North Am. 2002 Apr;33(2):359-66. doi: 10.1016/s0030-5898(01)00008-6. PMID 12389281
- [Background] Hong JY, Kim WS, Park J, Kim CH, Jang HD. Comparison of minimally invasive and open TLIF outcomes with more than seven years of follow-up. N Am Spine Soc J. 2022 Jun 11;11:100131. doi: 10.1016/j.xnsj.2022.100131. eCollection 2022 Sep. PMID 35783004
- [Background] Kleinert K, Theusinger OM, Nuernberg J, Werner CM. Alternative procedures for reducing allogeneic blood transfusion in elective orthopedic surgery. HSS J. 2010 Sep;6(2):190-8. doi: 10.1007/s11420-009-9151-6. Epub 2010 Jan 28. PMID 21886535
- [Background] Dodd RY. The risk of transfusion-transmitted infection. N Engl J Med. 1992 Aug 6;327(6):419-21. doi: 10.1056/NEJM199208063270610. No abstract available. PMID 1625717
- [Background] Myles PS, Smith JA, Forbes A, Silbert B, Jayarajah M, Painter T, Cooper DJ, Marasco S, McNeil J, Bussieres JS, McGuinness S, Byrne K, Chan MT, Landoni G, Wallace S; ATACAS Investigators of the ANZCA Clinical Trials Network. Tranexamic Acid in Patients Undergoing Coronary-Artery Surgery. N Engl J Med. 2017 Jan 12;376(2):136-148. doi: 10.1056/NEJMoa1606424. Epub 2016 Oct 23. PMID 27774838
- [Background] Danninger T, Memtsoudis SG. Tranexamic acid and orthopedic surgery-the search for the holy grail of blood conservation. Ann Transl Med. 2015 Apr;3(6):77. doi: 10.3978/j.issn.2305-5839.2015.01.25. No abstract available. PMID 25992376
- [Background] Badeaux J, Hawley D. A systematic review of the effectiveness of intravenous tranexamic acid administration in managing perioperative blood loss in patients undergoing spine surgery. J Perianesth Nurs. 2014 Dec;29(6):459-65. doi: 10.1016/j.jopan.2014.06.003. Epub 2014 Nov 20. PMID 25458625
- [Background] Xiong Z, Liu J, Yi P, Wang H, Tan M. Comparison of Intravenous versus Topical Tranexamic Acid in Nondeformity Spine Surgery: A Meta-Analysis. Biomed Res Int. 2020 Mar 9;2020:7403034. doi: 10.1155/2020/7403034. eCollection 2020. PMID 32219141
- [Background] Winter SF, Santaguida C, Wong J, Fehlings MG. Systemic and Topical Use of Tranexamic Acid in Spinal Surgery: A Systematic Review. Global Spine J. 2016 May;6(3):284-95. doi: 10.1055/s-0035-1563609. Epub 2015 Sep 21. PMID 27099820
- [Background] Gulabi D, Yuce Y, Erkal KH, Saglam N, Camur S. The combined administration of systemic and topical tranexamic acid for total hip arthroplasty: Is it better than systemic? Acta Orthop Traumatol Turc. 2019 Jul;53(4):297-300. doi: 10.1016/j.aott.2019.03.001. Epub 2019 Apr 4. PMID 30954338
- [Background] Li J, Wang L, Bai T, Liu Y, Huang Y. Combined use of intravenous and topical tranexamic acid efficiently reduces blood loss in patients aged over 60 operated with a 2-level lumbar fusion. J Orthop Surg Res. 2020 Aug 20;15(1):339. doi: 10.1186/s13018-020-01758-8. PMID 32819445
- [Background] Ker K, Edwards P, Perel P, Shakur H, Roberts I. Effect of tranexamic acid on surgical bleeding: systematic review and cumulative meta-analysis. BMJ. 2012 May 17;344:e3054. doi: 10.1136/bmj.e3054. PMID 22611164
- [Background] Murkin JM, Falter F, Granton J, Young B, Burt C, Chu M. High-dose tranexamic Acid is associated with nonischemic clinical seizures in cardiac surgical patients. Anesth Analg. 2010 Feb 1;110(2):350-3. doi: 10.1213/ANE.0b013e3181c92b23. Epub 2009 Dec 8. PMID 19996135
- [Background] Cravens GT, Brown MJ, Brown DR, Wass CT. Antifibrinolytic therapy use to mitigate blood loss during staged complex major spine surgery: Postoperative visual color changes after tranexamic acid administration. Anesthesiology. 2006 Dec;105(6):1274-6. doi: 10.1097/00000542-200612000-00029. No abstract available. PMID 17122592
- [Background] Murao S, Nakata H, Roberts I, Yamakawa K. Effect of tranexamic acid on thrombotic events and seizures in bleeding patients: a systematic review and meta-analysis. Crit Care. 2021 Nov 1;25(1):380. doi: 10.1186/s13054-021-03799-9. PMID 34724964
- [Background] Mikhail C, Pennington Z, Arnold PM, Brodke DS, Chapman JR, Chutkan N, Daubs MD, DeVine JG, Fehlings MG, Gelb DE, Ghobrial GM, Harrop JS, Hoelscher C, Jiang F, Knightly JJ, Kwon BK, Mroz TE, Nassr A, Riew KD, Sekhon LH, Smith JS, Traynelis VC, Wang JC, Weber MH, Wilson JR, Witiw CD, Sciubba DM, Cho SK. Minimizing Blood Loss in Spine Surgery. Global Spine J. 2020 Jan;10(1 Suppl):71S-83S. doi: 10.1177/2192568219868475. Epub 2020 Jan 6. PMID 31934525
- [Background] Montroy J, Hutton B, Moodley P, Fergusson NA, Cheng W, Tinmouth A, Lavallee LT, Fergusson DA, Breau RH. The efficacy and safety of topical tranexamic acid: A systematic review and meta-analysis. Transfus Med Rev. 2018 Feb 19:S0887-7963(17)30151-7. doi: 10.1016/j.tmrv.2018.02.003. Online ahead of print. PMID 29567052
- [Background] Mallepally AR, Mahajan R, Rustagi T, Goel SA, Das K, Chhabra HS. Use of Topical Tranexamic Acid to Reduce Blood Loss in Single-Level Transforaminal Lumbar Interbody Fusion. Asian Spine J. 2020 Oct;14(5):593-600. doi: 10.31616/asj.2019.0134. Epub 2020 Mar 30. PMID 32213797
- [Background] Wang F, Wang SG, Yang Q, Nan LP, Cai TC, Wu DS, Zhang L. Cytotoxicity and Effect of Topical Application of Tranexamic Acid on Human Fibroblast in Spine Surgery. World Neurosurg. 2021 Sep;153:e380-e391. doi: 10.1016/j.wneu.2021.06.125. Epub 2021 Jul 2. PMID 34224885
- [Background] Schwarzkopf R, Dang P, Luu M, Mozaffar T, Gupta R. Topical tranexamic Acid does not affect electrophysiologic or neurovascular sciatic nerve markers in an animal model. Clin Orthop Relat Res. 2015 Mar;473(3):1074-82. doi: 10.1007/s11999-014-4098-4. Epub 2015 Jan 6. PMID 25560955
- [Background] Ren Z, Li S, Sheng L, Zhuang Q, Li Z, Xu D, Chen X, Jiang P, Zhang X. Topical use of tranexamic acid can effectively decrease hidden blood loss during posterior lumbar spinal fusion surgery: A retrospective study. Medicine (Baltimore). 2017 Oct;96(42):e8233. doi: 10.1097/MD.0000000000008233. PMID 29049210
- [Background] Sudprasert W, Tanaviriyachai T, Choovongkomol K, Jongkittanakul S, Piyapromdee U. A Randomized Controlled Trial of Topical Application of Tranexamic Acid in Patients with Thoracolumbar Spine Trauma Undergoing Long-Segment Instrumented Posterior Spinal Fusion. Asian Spine J. 2019 Feb;13(1):146-154. doi: 10.31616/asj.2018.0125. Epub 2018 Oct 24. PMID 30347526
- [Background] Gybel M, Kristensen K, Roseva-Nielsen N. [Cardiac arrest caused by massive pulmonary embolism during treatment with tranexamic acid]. Ugeskr Laeger. 2013 May 13;175(20):1426-7. Danish. PMID 23663400
- [Background] Taparia M, Cordingley FT, Leahy MF. Pulmonary embolism associated with tranexamic acid in severe acquired haemophilia. Eur J Haematol. 2002 May;68(5):307-9. doi: 10.1034/j.1600-0609.2002.01607.x. PMID 12144537
- [Background] Krivokuca I, Lammers JW. Recurrent pulmonary embolism associated with a hemostatic drug: tranexamic acid. Clin Appl Thromb Hemost. 2011 Feb;17(1):106-7. doi: 10.1177/1076029609340902. Epub 2009 Oct 14. PMID 19833620
- [Background] Colomina MJ, Contreras L, Guilabert P, Koo M, M Ndez E, Sabate A. Clinical use of tranexamic acid: evidences and controversies. Braz J Anesthesiol. 2022 Nov-Dec;72(6):795-812. doi: 10.1016/j.bjane.2021.08.022. Epub 2021 Oct 7. PMID 34626756